CLINICAL TRIAL: NCT04512768
Title: Treating Comorbid Insomnia in Patients Receiving Transdiagnostic Internet-Delivered Cognitive Behaviour Therapy for Anxiety and Depression: A Randomized Controlled Trial
Brief Title: Treating Comorbid Insomnia in Transdiagnostic Internet-Delivered Cognitive Behaviour Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-204
Record Dates: First submitted 2020-08-04; First posted 2020-08-14 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Insomnia; Anxiety; Depression
Keywords: Internet-delivered Cognitive Behaviour Therapy; Insomnia; Depression; Anxiety; Transdiagnostic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard ICBT (Active Comparator): Participants in the Standard ICBT condition will receive an 8-week transdiagnostic course for anxiety and depression called The Wellbeing Course, originally developed by Macquarie University, Australia.
  Interventions: Behavioral: Transdiagnostic Internet-delivered Cognitive Behaviour Therapy
- Sleep-Enhanced ICBT (Experimental): Participants in the Sleep-Enhanced ICBT condition will receive an 8-week transdiagnostic course for anxiety and depression called The Wellbeing Course, originally developed by Macquarie University, Australia. In addition, participants in the Sleep-Enhanced ICBT condition will also receive a newly developed lesson designed to target insomnia.
  Interventions: Behavioral: Transdiagnostic Internet-delivered Cognitive Behaviour Therapy; Behavioral: Brief Internet-Delivered Cognitive Behaviour Therapy for Insomnia

INTERVENTIONS:
Behavioral: Transdiagnostic Internet-delivered Cognitive Behaviour Therapy — All participants receive an 8-week transdiagnostic course for anxiety and depression called The Wellbeing Course, originally developed by Macquarie University, Australia. The course is comprised of 5 lessons, beginning with psychoeducation and an introduction to the cognitive behavioural model, and then introducing key skills for managing anxiety and depression, including thought challenging, de-arousal strategies, graded exposure, behavioural activation, and relapse prevention. The course also includes supplementary resources that briefly provide information on related common concerns, such as managing worry, communication, assertiveness, problem solving, and a brief resource on sleep that provides limited psychoeducation and sleep hygiene information. Participants receive weekly brief therapist support via secure message or telephone from qualified counselors (social workers, psychologists).
Behavioral: Brief Internet-Delivered Cognitive Behaviour Therapy for Insomnia — A new sleep lesson will replace the existing resource, developed using a patient-oriented process, that provides information and skills to aid with insomnia. The sleep lesson includes psychoeducation on the nature of sleep problems and factors that affect sleep, such as circadian rhythm. Two key behavioural strategies are introduced: sleep restriction, which requires the patient to avoid napping and sleep on a strict schedule for several weeks until they begin to feel naturally sleepy at night; and stimulus control, which asks the participant to only spend time in bed when prepared to sleep and avoid other activities (e.g., work, TV) in bed. Patients will record how much they sleep each night and provide ratings of sleep quality and fatigue each week. Therapists will support patients in adjusting their sleep schedule. Patients are encouraged to apply skills they learn during the Wellbeing Course to sleep problems, for example, by applying thought challenging to beliefs about sleep.
  Arms: Sleep-Enhanced ICBT

SUMMARY:
Transdiagnostic Internet-delivered Cognitive Behaviour Therapy (ICBT) is an efficacious treatment option for anxiety and depression; however, not all patients benefit equally and some leave treatment before program completion. Comorbid symptoms of insomnia are extremely common among individuals seeking ICBT, yet sleep problems are rarely a primary focus of treatment in transdiagnostic ICBT despite insomnia being a known risk factor for anxiety and depression. This trial is designed to test whether an ICBT program for anxiety and depression can be improved by providing therapy for insomnia alongside the standard transdiagnostic program. For this randomized controlled trial, patients will be randomly assigned to receive either the standard ICBT program for anxiety and depression, which includes only brief supplementary information about sleep (n = 68), or a modified version that includes a lesson specifically on sleep (n = 132). The sleep lesson will introduce patients to two key behavioural strategies: sleep restriction and stimulus control, which previous research has demonstrated are effective at reducing insomnia. Patients will monitor their sleep throughout treatment and will complete measures of insomnia, anxiety and depression before treatment, at the end of the 8-week program, and 3 months after program conclusion to allow for a comparison of patient outcomes and completion rates between conditions. The acceptability of the new intervention will also be assessed by asking participants to provide feedback on the new materials and to complete measures of treatment satisfaction and working alliance.

ELIGIBILITY:
Inclusion Criteria:

* Participants must reside in Saskatchewan
* Participants must have access to a computer and feel comfortable using the internet
* Participants must be willing to provide a medical contact (e.g., family doctor) in case of medical emergency
* Participants must endorse some symptoms of anxiety or depression
* Participants must also endorse significant symptoms of insomnia (Insomnia Severity Index score of 10 or above)

Exclusion Criteria:

* High risk of suicide
* Unmanaged severe psychiatric illness (e.g., psychosis, mania)
* Severe alcohol or addictions problems that require referral
* High probability that another sleep disorder for which sleep restriction may be contraindicated is present (e.g., restless leg syndrome, sleep apnea, or sleep problems that are exclusively related to shift work)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Week 1 (pre-treatment), Week 8 (post-treatment), Week 20 (follow-up)
  Change in insomnia symptoms from pre-treatment (Week 1) to post-treatment (8 weeks) and from pre-treatment to follow-up (20 weeks). The ISI is a brief measure of insomnia comprised of 7 questions that ask about difficulties falling asleep, staying asleep, and waking too early, which respondents answer on a scale from 0 (None) to 4 (Very Severe), producing a score between 0 and 28.
Patient Health Questionnaire 9-item (PHQ-9) | Week 1 (pre-treatment), Week 8 (post-treatment), Week 20 (follow-up)
  Change in depression symptoms from pre-treatment (Week 1) to post-treatment (8 weeks) and from pre-treatment to follow-up (20 weeks). The PHQ-9 is a 9-item self-report measure of symptoms of depression that produces a total depression severity score ranging from 0-27.
Generalized Anxiety Disorder (GAD-7) | Week 1 (pre-treatment), Week 8 (post-treatment), Week 20 (follow-up)
  Change in anxiety symptom from pre-treatment (Week 1) to post-treatment (8 weeks) and from pre-treatment to follow-up (20 weeks). The GAD-7 is a 7-item self-report measure of symptoms of anxiety that produces a total anxiety severity score ranging from 0-21.

SECONDARY OUTCOMES:
Panic Disorder Severity Scale (PDSS) | Week 1 (pre-treatment), Week 8 (post-treatment), Week 20 (follow-up)
  Change in symptoms of panic. The PDSS is a 7-item measure of common symptoms of panic disorder. Respondents answer each item on a 0-4 scale, producing a total score between 0 and 28.
Social Interaction Anxiety Scale and Social Phobia Scale - Short Form (SIAS-6/SPS-6) | Week 1 (pre-treatment), Week 8 (post-treatment), Week 20 (follow-up)
  Change in symptoms of social anxiety. The SIAS-6/SPS-6 includes 12 items related to common symptoms of social anxiety that are summed to create a total score.
Treatment Satisfaction | Week 8 (post-treatment)
  A treatment satisfaction questionnaire that includes questions about the patient's opinion of the program and the working alliance they developed with their therapist. Patients will also be asked whether they would recommend the treatment to others. Patients will then complete the Working Alliance Inventory-Short a 12-item measure of the therapeutic alliance.
Lesson Completion | Ongoing throughout treatment (Weeks 1-8)
  The program website will record when patients access each lesson, providing a way to calculate the proportion of patients who complete each lesson and treatment overall.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Edmonds, MA, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
Other researchers may ask to review IPD from this trial following completion of data collection. For the purposes of meta-analyses or other legitimate uses, IPD will be provided after being fully de-identified.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available for a period beginning 6 months after the conclusion of the trial until 5 years have elapsed.
Access Criteria: Data will be provided to researchers who provide a methodologically sound proposal and present a request for data that is within our operational capacity to provide. Additionally, researchers must provide information about how they will use and store the data, as well as sign an agreement related to the use of the data.